CLINICAL TRIAL: NCT06684769
Title: Non-surgical Treatment of Mandibular and Maxillary Molar Furcations With a Chitosan Brush With Adjunct Enamel Matrix Derivative- a Split-mouth Randomized Clinical Trial
Brief Title: A Chitosan Brush and Enamel Matrix Derivative for Non-surgical Treatment of Furcations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riga Stradins University (Other)
Collaborators: University of Turku (Other); University of Oslo (Other); Labrida AS (Industry)
Responsible Party: Principal Investigator, Anete Vaškevica, Lectureur, Riga Stradins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-PĒK-4/659/2024
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Periodontitis, Adult; Furcation Defects; Furcation of Root of Tooth; Periodontitis Complex
MeSH Terms: conditions — Chronic Periodontitis; Furcation Defects

STUDY DESIGN:
Intervention Model Description: Randomised, single-blinded, split-mouth clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chitosan brush with Emdogain FL (Experimental): Furcation Involved areas will be treated with the oscillating chitosan brush Labrida BioClean® and Straumann® Emdogain® FL at Baseline
  Interventions: Device: Emdogain® FL; Device: Labrida BioClean®
- Chitosan brush alone (Sham Comparator): Furcation Involved areas will be treated with the oscillating chitosan brush Labrida BioClean® at Baseline
  Interventions: Device: Labrida BioClean®

INTERVENTIONS:
Device: Emdogain® FL — Enamel Matrix Derivatives
  Arms: Chitosan brush with Emdogain FL
Device: Labrida BioClean® — Oscillating Chitosan Brush

SUMMARY:
Patients diagnosed with stage III or IV periodontitis who exhibit mandibular first or second molars with Class II, Subclass A, or B buccal and/or lingual mandibular furcation defects (horizontal probing depth of ≥ 3 mm ) will be recruited.

Patients diagnosed with stage III or IV periodontitis who exhibit maxillary first or second molars with Class II, Subclass A, or B buccal furcation defects (horizontal probing depth of ≥ 3 mm ) if furcation involvement on the palatal side (mesiopalatal and distopalatal) does not exceed Class 1 will be recruited.

This study will be a prospective, randomized, single-blinded, controlled clinical trial with a split-mouth design.

Patients will be recruited from the clinics of the Riga Stradiņš University Institute of Stomatology of Riga, Latvia.

Before the baseline treatment, all patients who meet the inclusion criteria will be given detailed oral hygiene instructions and motivation.

Patients' furcation defects in each quadrant will be randomly allocated at a 1:1 ratio to either the application of Oscillating Chitosan Brush with Enamel Matrix Derivatives (test group) or Oscillating Chitosan Brush alone (control group).

Non-surgical periodontal treatment of furcation defects on the test side will be performed through the application of Oscillating Chitosan Brush with Enamel Matrix Derivatives and on the control side with Oscillating Chitosan Brush alone.

The re-evaluation of periodontal status will be performed 12 weeks following the baseline treatment.

Biofilm samples and gingival crevicular fluid (GCF) samples will be taken at the baseline and at 4 weeks.

ELIGIBILITY:
Inclusion criteria:

1. The patient is 18 years of age or older
2. The patient does not have any systemic diseases that may affect the results of the study
3. The patient has a plaque index of 20% or less at the study entry
4. The patient has a history of severe localized or generalized periodontitis (stage III or IV)
5. Completed the first and second steps of periodontal treatment (According to Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline) (Sanz M. et al.)
6. Buccal and/or lingual Class 2A and/or 2B furcation involvement (FI) defects on both sides of the Mandibular first and/or second molars after completing the first and second steps of periodontal treatment.
7. Buccal Class 2A and/or 2B furcation involvement (FI) defects on both sides of the maxillary first and/or second molars after completion of the first and second step of periodontal treatment if furcation involvement on the palatal side (mesiopalatal and distopalatal) does not exceed Class 1.
8. Psychological appropriateness
9. Consents to all follow-up visits

Exclusion Criteria:

1. Patients who have systemic diseases that may affect the results of the study
2. Use of medications that may affect study results (anti-osteoporotic drugs, statins, corticosteroids, anticoagulants)
3. Patients who use calcium channel blockers, cyclosporine A or antiepileptic drugs if there are clinically visible hyperplastic changes in the gingival margin.
4. Patients who have received any type of systemic antibiotics in the last six months prior to the start of the study and patients starting antibiotics during the study
5. Patients requiring antibiotic premedication prior to periodontal treatment
6. Oncological disease
7. Chemotherapy and/or radiotherapy (active or history)
8. Pregnancy and breastfeeding
9. Any condition or current treatment which, in the opinion of the investigator and/or consulting physician, may present an unreasonable risk
10. Psychoemotional disorders and depression
11. Use of antipsychotic medication or antidepressants
12. Lack of patient motivation to undertake adequate dental care at home or complete periodontal treatment, patients residing outside Latvia
13. Molars with combined endodontic-periodontal lesions, active endodontic infection
14. Prosthetic factors for molars not allowing clinical measurements
15. Huge restoration or amalgam fillings that could potentially cause fractures or furcation involvement
16. Enamel pearls or filling or crown margins
17. Decay or root resorption
18. Tooth mobility degree 3
19. Molars in which the gingival margin is positioned apically from the entrance into the furcation area
20. Clinical attachment level and or pockets mesial and distal to the furcation involvement defect of 6 or more mm
21. Strong vomiting reflex that would prevent adequate periodontal treatment
22. People close to the study subjects, work colleagues, relatives, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Modified Bleeding on Probing index (mBoP) | Baseline, 12 weeks
  Pseudo marker of inflammation, lower scores mean a better outcome 0 = no bleeding;
  1. = a bleeding spot;
  2. = a bleeding line;
  3. = pronounced bleeding within 30 seconds following probing of the pocket
Probing Pocket Depth (PPD) in mm | Baseline,12 weeks
  Pseudo marker of inflammation, lower scores mean a better outcome.
Clinical Attachment Level (CAL) in mm | Baseline, 12 weeks
  Marker of gain in attachment, lower scores mean a better outcome
Furcation Involvement 1 | Baseline, 12 weeks
  Marker of gain in attachment, Horizontal Furcation involvement measurement using Nabers Probe
  1. Horizontal loss of periodontal tissue support less than 3 mm
  2. Horizontal loss of support 3 mm or more, but not encompassing the total width of the furcation
  3. Horizontal through-and-through destruction of the periodontal tissue in the furcation Lower scores mean a better outcome
Furcation Involvement 2 in mm | Baseline, 12 weeks
  Marker of gain in attachment, Horizontal Furcation involvement measurement using UNC 15mm probe, lower scores mean a better outcome

SECONDARY OUTCOMES:
Proteomic profile of gingival crevicular fluid (GCF) | Baseline, 4 weeks,
  Differences in the GCF of regeneration-related marker concentrations between test and control groups
Microbiological changes in microbial plaque | Baseline, 4 weeks,
  Differences in the microbial profile between test and control groups
Visual analog scale (VAS) | Baseline
  Evaluation of self-perceived pain using a 100 mm Visual analog scale (range 0 - 100) at baseline treatment visit; 0 - no pain, 100 - worst pain ever felt. Lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ilze Akota, PhD, Study Chair — Riga Stradins University
Locations (1):
- Riga Stradins University Institute of Stomatology, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No